CLINICAL TRIAL: NCT06054607
Title: Effect of Short-chain Fatty Acids on Aerobic Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 23-13H; M-11031 (Other: HQ US Army Medical Research and Development Command IRBO)
Record Dates: First submitted 2023-08-21; First posted 2023-09-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Aerobic Endurance; Metabolism
Keywords: short-chain fatty acid; microbiome; endurance; fiber; resistant starch; gastrointestinal
MeSH Terms: interventions — Butyrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-amylose maize starch (Placebo Comparator): Low-amylose maize starch (AMIOCA; Ingredion, Inc).
  Interventions: Other: Low-amylose maize starch
- High-amylose maize starch+acetate/butyrate (Active Comparator): High-amylose maize starch, (Hylon VII; Ingredion, Inc.) to which the SCFA acetate or butyrate has been chemically added.
  Interventions: Dietary Supplement: High-amylose maize starch+acetate/butyrate

INTERVENTIONS:
Dietary Supplement: High-amylose maize starch+acetate/butyrate — High-amylose maize starch (HAMS), commercially available as Hylon VII (Ingredion, Inc.), to which the SCFA acetate or butyrate has been chemically added. Hylon VII is a HAMS containing ~70% amylose and used in a variety of food products. To produce SCFA-enriched HAMS, Hylon VII is chemically modified through esterification with the SCFA acetate or butyrate.
  Arms: High-amylose maize starch+acetate/butyrate
Other: Low-amylose maize starch — Rapidly digestible low-amylose maize starch (0% amylose, 100% amylopectin) sold commercially as AMIOCA (Ingredion, Inc).
  Arms: Low-amylose maize starch

SUMMARY:
Randomized, double-blind, placebo-controlled crossover study designed to determine the effects of increasing colonic short-chain fatty acid (SCFA) content on aerobic endurance in healthy adults, and to identify underpinning mechanisms. In random order, healthy physically active adults will consume provided diets low in fiber and supplemented with SCFA-enriched high amylose maize starch (a poorly digested resistant starch considered a fermentable fiber) or low amylose maize starch (a rapidly digestible starch) for 1-week separated by a ≥2-week washout. At the end of each intervention period, participants will complete an endurance exercise bout followed by a time trial. Biological samples will be collected to assess muscle and whole body metabolism, gut microbiota, inflammation, and gastrointestinal function.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 39 years (active-duty personnel who are 17 yr of age will also be allowed to participate).
* In good health.
* Routinely participate in moderate or higher intensity aerobic and/or resistance exercise at least 4 days per week for ≥20 min/d.
* Meet Army weight for height and body composition standards as defined in Army Regulation 600-9.
* Self-reports a usual bowel movement frequency of every other day or more often.
* Willing to refrain from the use of caffeine, alcohol, and nicotine while consuming study diets.
* Willing to refrain from all dietary supplements beginning 2 weeks prior to study start and throughout study participation.
* Willing to refrain from consumption of any foods containing live microorganisms (e.g., yogurt, kefir, kombucha) or added prebiotics (e.g. Fiber One products) beginning 2 weeks prior to study start and throughout study participation.
* Willing to participate in all study procedures.
* Females must have normal menstrual cycles between 26-32 days in duration; 5 menstrual cycles within the past 6 months; or be using an oral/hormonal contraceptive which contains low-dose estrogen/progesterone to maintain continuous levels throughout the 28-day cycle (i.e., no placebos).

Exclusion Criteria:

* Females who are pregnant, expecting to become pregnant during the study, or breastfeeding.
* Any of the following medical conditions:

Cardiac disease (including arrhythmia or fast or skipped heart beats) Hypertension Musculoskeletal injuries that compromise exercise capability Metabolic or cardiovascular abnormalities (e.g., kidney disease, diabetes, etc.) Disease of the GI tract including, but not limited to diverticulitis, inflammatory bowel disease, irritable bowel syndrome, peptic ulcer disease, Crohn's disease, and ulcerative colitis Allergy to skin adhesive or Lidocaine (or other local anesthetic being used in place of Lidocaine) Suspected or known strictures, fistulas, or physiological/mechanical GI obstruction History of gastric bezoar Swallowing disorders; severe dysphagia to food or pills Implanted or portable electro-mechanical medical devices (e.g., pacemaker)

* Colonoscopy within 3 months of study participation.
* Any use of antibiotics or antimycotics, except topical antibiotics/antimycotics, within 3 months of study participation.
* Regular (i.e., weekly or more frequent) use of over-the-counter medications (including antacids, laxatives, stool softeners, and anti-diarrheals) unless approved by study PI.
* Use of medication (i.e., diabetes medications, statins, corticosteroids, etc.) that affects macronutrient utilization and/or the ability to participate in strenuous exercise.
* Anemia (HCT <38 for men and <34 for women) or Sickle Cell Anemia/Trait.
* Not willing or able to follow all study procedures and diet/exercise restrictions.
* Allergies, intolerances, unwillingness or inability to eat provided foods and beverages.
* Following vegetarian/vegan diet or other highly restrictive diet (e.g., ketogenic diet, very high protein diet, Paleo diet, etc.).
* Any previous blood donation within the previous 8 weeks that when combined with the volume of blood collected for the study within any 8-week period would exceed 550mL.

Ages: 17 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Run time | Phases 1 and 2, day 8
  Time to complete a 5km treadmill run

SECONDARY OUTCOMES:
Muscle glycogen content | Phases 1 and 2, day 8
  Muscle glycogen content
Plasma glucose turnover | Phases 1 and 2, day 8
  Glucose production, utilization and metabolic clearance rate measured during endurance steady state exercise using 6,6-[2H2] glucose tracer
Whole body substrate oxidation | Phase 1 and 2, day 8
  Carbohydrate and fat oxidation rates measured during endurance steady state exercise using indirect calorimetry
Serum short-chain fatty acid concentrations | Phases 1 and 2, day 8. Measured fasted (-300 minutes) and before (0 minutes) and at the end (80 minutes) of steady state endurance exercise
  Serum acetate, butyrate and propionate concentrations
Fecal short-chain fatty acid concentrations | Phases 1 and 2, days 1 and 7
  Fecal acetate, butyrate and propionate concentrations
Intestinal permeability | Phases 1 and 2, day 8
  Small and large intestine permeability measured by saccharide excretion in urine

OTHER OUTCOMES:
Gastrointestinal symptoms | Phases 1 and 2, daily on days 1 through 8
  Gastrointestinal symptoms (bloating, pain, nausea, flatulence, discomfort, urge to defecate) measured by 10 cm (0 = low, 10 = high) visual analog scale
Circulating biomarkers of substrate utilization | Phases 1 and 2, day 8. Measured before (-300minutes, 0minutes) and during (20, 40, 60, 80minutes) steady state endurance exercise.
  Serum/plasma glucose, insulin, free fatty acids, glycerol, lactate and beta-hydroxybutyrate
Total protein content in muscle | Phases 1 and 2, day 8
  Total protein content measured in muscle collected before and after steady state endurance exercise.
Total protein expression of molecular markers associated with regulation of muscle metabolism. | Phases 1 and 2, day 8
  Muscle protein signalling measured by Western blotting in muscle collected before and after steady state endurance exercise. Total protein expression of molecular markers associated with regulation of muscle metabolism will be measured to include (but not be limited to): Akt, p-AktSer473, AMPKα, p- AMPKαThr172, PGC-1α , SIRT1, ACC, p-ACCSer79, p53, p-p53Ser15, PDK4, IRS1, p-IRS1Ser302, GSK-3β, p-GSK-3βSer9, GSK-3α , p-GSK-3α Ser21, GS, p-GSSer641, and GLUT4.
Phosphorylation status of molecular markers associated with regulation of muscle metabolism. | Phases 1 and 2, day 8
  Muscle protein signalling measured by Western blotting in muscle collected before and after steady state endurance exercise. Phosphorylation status of molecular markers associated with regulation of muscle metabolism will be measured to include (but not be limited to): Akt, p-AktSer473, AMPKα, p- AMPKαThr172, PGC-1α , SIRT1, ACC, p-ACCSer79, p53, p-p53Ser15, PDK4, IRS1, p-IRS1Ser302, GSK-3β, p-GSK-3βSer9, GSK-3α , p-GSK-3α Ser21, GS, p-GSSer641, and GLUT4 .
Pyruvate dehydrogenase activity in muscle | Phases 1 and 2, day 8
  Pyruvate dehydrogenase activity in muscle before and after steady state endurance exercise measured colorimetric assay.
Gene expression | Phases 1 and 2, day 8
  Expression of genes regulating carbohydrate and fat oxidation in muscle collected before and after steady state endurance exercise. Individual primers will be used to determine the mRNA expression of known intracellular targets regulating substrate metabolism to include (but not limited to): FAT, PDK4, HADHA, PGC-1α, PPARδ, PPARγ, FABP, CPT1a, ACOX1, GS, GSK3α, GLUT4, and HK2.
microRNA expression | Phases 1 and 2, day 8
  Expression of genes and microRNA regulating carbohydrate and fat oxidation in muscle collected before and after steady state endurance exercise. microRNA analysis will be conducted using microarray, assessing microRNA that may be associated with substrate metabolism.
Gut microbiota composition | Phases 1 and 2, days 1 and 7
  Relative abundance of bacterial taxa measured by 16S rRNA amplicon sequencing
Gut microbiome gene content | Phases 1 and 2, days 1 and 7
  Relative abundances of microbial genes measured by shotgun metagenomics sequencing
Circulating biomarkers of inflammation | Phases 1 and 2, day 8. Measured before (-300minutes) and at the end (80minutes) of steady state endurance exercise.
  Serum interleukin (IL)-6, IL-10, IL-17, IL-8, IL-1ralpha, IL-1beta, tumor necrosis factor-alpha, interferon gamma
Circulating biomarkers of gut barrier function | Phases 1 and 2, day 8. Measured fasted (-300minutes) and before (0minutes), during (40minutes) and at the end (80minutes) of steady state endurance exercise.
  Serum claudin-3, intestinal fatty acid binding protein and zonulin
Circulating microRNA | Phases 1 and 2, day 8. Measured fasted (-15minutes) and at the end (80minutes) of steady state endurance exercise.
  Serum C-microRNA
Appetite | Phases 1 and 2, daily on days 1 through 7
  Appetite (hunger, fullness, desire to eat, prospective consumption) measured by 10 cm (0 = low, 10 = high) visual analog scale
Breath hydrogen and methane | Phases 1 and 2, day 8. Measured fasting (-300minutes) and before (0minutes) and at the end (80minutes) of steady state endurance exercise
  Breath hydrogen and methane concentrations

CONTACTS AND LOCATIONS:
Overall Officials: J. Philip Karl, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- United States Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data and samples will remain under the control of the Principal Investigator and may be shared with outside collaborators for future research with appropriate data sharing agreements and legal/ethical approvals. De-identified microbiome sequencing data may be posted in a publicly available data repository.

DOCUMENTS (1):
  • Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT06054607/ICF_000.pdf